CLINICAL TRIAL: NCT03081975
Title: Comparison of Adenoma Detection Rate Using Narrow Band Imaging Versus HD White Light Colonoscopy in Screening and Surveillance Colonoscopies
Brief Title: Comparison of ADR Using NBI Versus HD White Light Colonoscopy in Screening and Surveillance Colonoscopies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jena University Hospital (Other)
Responsible Party: Principal Investigator, Martin Bürger, Narrow band imaging does not increase adenoma detection rate compared to high definition white light colonoscopy in screening and surveillance colonoscopies, Jena University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: NBI01
Record Dates: First submitted 2017-03-04; First posted 2017-03-17 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Narrow Band Imaging
Keywords: adenoma detection rate; narrow band imaging
MeSH Terms: interventions — Narrow Band Imaging

ARMS (2):
- HD white light (Active Comparator): Colonoscopy was performed by use of HD-WLC or HD-NBI upon withdrawal
  Interventions: Device: HD white light or NBI
- HD narrow band imaging (Active Comparator): Colonoscopy was performed by use of HD-WLC or HD-NBI upon withdrawal
  Interventions: Device: HD white light or NBI

INTERVENTIONS:
Device: HD white light or NBI — Use of NBI or HD white light

SUMMARY:
The aim of this study is to compare ADR using HD-NBI or HD-WLE during screening and surveillance colonoscopies.

DETAILED DESCRIPTION:
Background:

Despite recent advances in endoscopic technology adenoma miss rate still is up to 20% and contributes to the occurrence of interval cancers. Therefore, improved imaging modalities have been introduced to increase adenoma detection rate (ADR) during screening and surveillance colonoscopies. Recently, narrow band imaging (NBI; Exera II series, Olympus Corporation) was not significantly better than high definition white light colonoscopy (WLC) for the detection of patients with colorectal polyps, or colorectal adenomas1. However, Olympus' current Exera III series is characterized by better illumination of the bowel lumen and may be associated with a higher ADR than high definition WLC.

Methods:

Investigators performed a prospective evaluation in patients referred to the Department of Interdisciplinary Endoscopy at Jena University Hospital for screening or surveillance colonoscopy between January and November 2015 in daily clinical practice. Colonoscopy was performed by use of HD-WLC or HD-NBI upon withdrawal of the colonoscope (Exera III series, Olympus Corporation).

ELIGIBILITY:
Inclusion Criteria:

* Screening colonoscopies

Exclusion Criteria:

* Insufficient bowel cleansing
* Age under 55years

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2015-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Adenoma detection rate | up to 60min
  Adenoma detection rate

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Schmidt, MD, Study Director — University Clinic Jena
Locations (1):
- University Clinic Jena, Jena, Thueringia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Burger M, Weber M, Petersen I, Stallmach A, Schmidt C. Adenoma detection rate using narrow-band imaging is inferior to high-definition white light colonoscopy in screening and surveillance colonoscopies in daily clinical care: A randomized controlled trial. Medicine (Baltimore). 2022 Aug 12;101(32):e29858. doi: 10.1097/MD.0000000000029858. PMID 35960070